CLINICAL TRIAL: NCT03442023
Title: Differences Between Oral Colonization Rates of Gram-negative Bacteria in ICU Patients When Using Chlorhexidine Mouthwash at 0.12% Versus Chlorhexidine Mouthwash at 2.0%
Brief Title: Different Oral Colonization of Gram-negative Bacteria in ICU Patients When Using Chlorhexidine at 0.12% Versus Chlorhexidine at 2.0%
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Guanajuato (Other)
Responsible Party: Principal Investigator, Jose Antonio de Jesus Alvarez Canales, PhD, MD, MSCR, Universidad de Guanajuato
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSGTO00153
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Chlorhexidine; Ventilator Associated Pneumonia
Keywords: Chlorhexidine; Gram-negative; Colonization
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlorhexidine 2% (Experimental): Subjects in this arm will receive standard care plus mouth rinse every 12 hours via spray with 2% chlorhexidine concentration, one week intervention, Drug: Chlorhexidine gluconate at 2%
  Interventions: Drug: Chlorhexidine gluconate at 2%
- Chlorhexidine 0.12% (Active Comparator): Subjects in this arm will receive standard care plus mouth rinse every 12 hours via spray with 0.12% chlorhexidine concentration, one week intervention, Drug: Chlorhexidine gluconate at 0.12%
  Interventions: Drug: Chlorhexidine gluconate at 0.12%

INTERVENTIONS:
Drug: Chlorhexidine gluconate at 2% — Mouth Rinse with Chlorhexidine gluconate at 2% every 12 hours, one week.
  Arms: Chlorhexidine 2%
Drug: Chlorhexidine gluconate at 0.12% — Mouth Rinse with Chlorhexidine gluconate at 0.12% every 12 hours, one week.
  Arms: Chlorhexidine 0.12%

SUMMARY:
This study will assess the utility of different chlorhexidine mouthwash concentrations on ICU patients to decolonize their oral cavities from gram-negative bacteria, since this is a non-desirable condition that leads to higher mortality rates and longer hospitalization times. One group will receive the 0.12% chlorhexidine mouthwash and the other group will receive the 2% chlorhexidine mouthwash.

ELIGIBILITY:
Inclusion Criteria:

* Patients with minimum required age of consent that were admitted to the intensive care unit and who received at least 48 hours of mechanical ventilation.

Exclusion Criteria:

* Patients who wish to withdraw consent and leave the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Gram-negative decolonization rate | 2 weeks
  Patients admitted to the ICU who were originally colonized with gram-negative bacteria and at the end of the study are no longer colonized by gram-negative bacteria.
Gram-negative colonization rate | 2 weeks
  Patients admitted to the ICU who were originally not colonized with gram-negative bacteria and at the end of the study are colonized by gram-negative bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Alvarez, PhD, Principal Investigator — Universidad de Guanajuato
Locations (1):
- University of Guanajuato, León, Guanajuato, Mexico